CLINICAL TRIAL: NCT06412315
Title: The Effects of Citalopram on the Brain's Response to Faces
Brief Title: 7T Amygdala and Citalopram Study
Acronym: 7TAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Catherine Harmer, Professor of Cognitive Neuroscience, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7T_Amygdala_Citalopram
Record Dates: First submitted 2024-03-01; First posted 2024-05-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Emotional Processing; Cognition; Mood Disorders; Depressive Disorder; Depression
Keywords: Antidepressants; Experimental medicine; Psychopharmacology; Emotional Processing; fMRI; High field strength fMRI; 7 Tesla MRI
MeSH Terms: conditions — Mood Disorders; Depressive Disorder; Depression | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive citalopram or placebo. Citalopram is not being administered for treatment purposes, the purpose is to understand the mechanisms underpinning its effects (no clinical outcome measure).
  A double-blind randomised placebo-controlled design (25 participants in each group) will be used, with 1 single dose of citalopram (20mg) or placebo.
Who Masked: Participant, Investigator
Masking Description: All members of the study team will be blinded to the condition a participant is allocated to with the exception of the team member responsible for treatment allocation (who will not interact with the participant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram (Experimental)
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Participants will receive a single dose (20mg) citalopram. Tablets encapsulated to aid blinding. To take per oral once.
  Arms: Citalopram
Drug: Placebo — Participants will receive a single dose of placebo (sucrose). Tablets encapsulated to aid blinding. To take per oral once
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate how a common antidepressant citalopram (which increases the levels of the chemical messenger serotonin), affects how a key area of the brain involved in depression (the amygdala) responds to emotional information.

Healthy participants will undergo medical and psychiatric health screening, after which they will be assigned to receive either a single dose of citalopram (20mg) or placebo, and undergo brain scanning (7T fMRI) whilst viewing emotional faces. Since the scan uses high field strength, the investigators will be able to see effects of citalopram on different subfields within the amygdala which will help to understand how citalopram might be working.

DETAILED DESCRIPTION:
Antidepressants typically decrease amygdala response to negative stimuli while enhancing response to positive stimuli, but it is unclear at a mechanistic level how increasing serotonin would have this opposing effect. One hypothesis is that although positive and negative cues activate the same area at a global level, more detailed characterisation may reveal key differences in processing in terms of localisation or response function. Until now, due to methodological restriction, the amygdala has been mostly studied as a single structure. It is however known that it consists of a number of subfields, which are likely to play distinct roles in emotional processing. In this study the investigators will make use of 7T fMRI scanning to study the effects of a single dose (20 mg) of citalopram (selective serotonin reuptake inhibitor, SSRI) on these subfields during emotional face processing, allowing greater precision to identify underlying neural mechanisms underpinning psychological effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Sufficiently fluent English to understand and complete the task

Exclusion Criteria:

* Participants with ferromagnetic objects in their bodies (e.g. metal implants, vessel clips, shrapnel injuries) or with implanted devices which may be damaged by the magnet (e.g. heart pacemakers)
* Any other MRI contraindication following MRI safety screening
* History or current significant psychiatric illness (like major depressive disorder)
* Current or past diagnosis of any significant personality disorder (e.g. borderline personality disorder) according to self-report
* Diagnosis of attention deficit hyperactive disorder or autistic spectrum disorder that impairs daily functioning, requires pharmacotherapy or in the opinion of the study medic would affect the scientific integrity of the study
* Currently or within last 3 months taking psychoactive medications (requires further discussion with researcher)
* Current or within the last 3 months use of medication that might interact with the effects of citalopram or affect the scientific integrity of the study
* Known contraindication to citalopram including: past allergic reaction to citalopram or any other medicines, diagnosis of a cardiovascular condition, glaucoma, type 1 or type 2 diabetes, diagnosis of epilepsy, previous diagnosis of angle-closure glaucoma, or current use of any other medication whose use interacts with citalopram (according to British National Formulary (BNF) guidance) e.g. associated with prolonged QT-interval
* Any other current or past medical conditions which in the opinion of the study medic may interfere with the safety of the participant or the scientific integrity of the study including epilepsy/seizures, brain injury, hepatic or renal disease, diabetes, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, neurological conditions
* Clinically significant abnormal values for urine drug screen, pulse, and blood pressure measurement (in accordance with Best Practice Guidance 13: 'Non-invasive measurement of blood pressure'). A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Current alcohol or substance misuse disorder
* Body Mass Index under 18 and over 30
* Pregnant or planning a pregnancy, or breast feeding
* Previously taken part in a study that used similar computer tasks (MRI faces task, emotional test battery) as those in the present study
* Participation in a study that involves the use of a psychoactive medication or brain stimulation within the last three months
* Use of recreational drugs (e.g. cannabis, cocaine, amphetamines) within last three months
* Smoking > 5 cigarettes per day, or vape a comparable amount (> 0.5ml / a quarter of a 2ml vape);
* Typically drinks > 6 caffeinated drinks per day (e.g. tea, coffee, coca cola, Red Bull)
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Neural measures: fMRI BOLD univariate analysis | 3 hours after dosing for approximately 1 hour
  Blood-oxygen-level-dependent (BOLD) fMRI (region of interest (ROI) analysis amygdala) during the performance of an emotional faces task.
  Differential amygdala response to fearful and happy faces.
  Univariate analysis
Neural measures: fMRI BOLD multivariate analysis | 3 hours after dosing for approximately 1 hour
  Blood-oxygen-level-dependent (BOLD) fMRI (region of interest (ROI) analysis amygdala) during the performance of an emotional faces task.
  Amygdala response to fearful and happy faces. Multivariate pattern analysis.

SECONDARY OUTCOMES:
Behavioural measures: Accuracy during gender discrimination task | 3 hours after dosing for approximately 1hour
  Accuracy (% correct) of gender identification will be measured to ensure participant engagement throughout the task.
Behavioural measures: Reaction times during gender discrimination task | 3 hours after dosing for approximately 1hour
  Reaction times (ms) of gender identification will be measured to ensure participant engagement throughout the task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Department of Psychiatry, Oxford, Oxfordshire, United Kingdom